CLINICAL TRIAL: NCT05544877
Title: An Energetic View on Creativity, Psychopathology and Intelligence: A Mixed Design Study in Adults With and Without Psychological Disorders
Brief Title: An Energetic View on Creativity, Psychopathology and Intelligence: The Brain2Business Study
Acronym: B2B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Psychiatrische Dienste Thurgau (Other)
Collaborators: Brain2Go AG (Unknown); greenTEG AG (Industry); SOMNOmedics GmbH (Unknown)
Responsible Party: Principal Investigator, Rainer Krähenmann, Medical director of Psychiatric Services Thurgau (PD Dr.), Psychiatrische Dienste Thurgau
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PDT_024_B2B
Record Dates: First submitted 2022-07-30; First posted 2022-09-19 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: General Psychopathology; Fatigue; Depressive Disorder, Major
Keywords: General psychopathology; Fatigue; Depression; somatoform disorders; Internalizing disorders; Thought disorders; Detachment disorders; Disinhibited externalizing disorders; Antagonistic externalizing disorders; Behavioral Activation; Gratefulness exercise; Creativity technique; Brain2Business; Solo Brainstorming
MeSH Terms: conditions — Fatigue; Depressive Disorder, Major; Depression; Somatoform Disorders

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned in blocks of 20 and stratified for psychological disorder (with/without self-reported lifetime or current diagnosis of a psychological disorder) to one of two creativity technique conditions (Brain2Business vs Solo Brainstorming).
Who Masked: Participant
Masking Description: Based on the behavioral intervention, the administrator of the intervention who is intrinsically also the outcome assessor of the primary outcome cannot be masked. Participants are masked as they are not aware about their treatment condition. Self-rated questionnaire-based outcome measures are not subject to bias as participants are masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brain2Business (B2B) (Experimental): The Brain2Business (B2B) technique aims to improve creative thinking. It is a game-based "conceptual combination" method that is performed by the participant with support of one trained B2B administrator in a laboratory session and without support in 5 at-home sessions. In this technique, thirty-six different images are randomly selected on a board by throwing two dices. Inspired by these images, participants are asked to create new ideas regarding three questions for a total of at least 39 minutes over a period of 5 days. One question is from a standardized creativity test and two questions are part of psychotherapeutic techniques (idea generation for pleasurable activities within behavioral activation (PA-BA) and for a gratefulness exercise (GE)). The B2B technique is based on the principles of solo brainstorming (SBS). A trained B2B administrator is documenting the answers of the participant, and mentioning the principles of SBS (see SBS group).
  Interventions: Behavioral: Integrated 5-day Gratitude Exercise and Behavioral Activation Program
- Solo Brainstorming (SBS) (Active Comparator): Solo brain storming (SBS) is the active control condition. The technique aims to improve creative thinking through the principles of SBS. SBS principles include i) idea quantity goes before quality, ii) no criticism and evaluation of ideas during idea generation, iii) original ideas are encouraged. The principles are provided to participants in the same way, with the same questions to be answered, and over the same time period as in the B2B group. A trained SBS administrator is documenting the answers of the participant, and mentioning the principles of SBS.
  Interventions: Behavioral: Integrated 5-day Gratitude Exercise and Behavioral Activation Program

INTERVENTIONS:
Behavioral: Integrated 5-day Gratitude Exercise and Behavioral Activation Program — The 5-day intervention integrates a brief behavioral activation (BA) and a gratefulness exercise (GE) program. BA is composed of a lab-based idea generation and planning phase as well as a home-based performing phase with regard to pleasurable activities. GE is a idea generation task about aspects in life participants are grateful for about. It is performed once lab-based and daily with a home-based diary.

SUMMARY:
The interventional part of the study aims to assess the acute effect of the Brain2Business (B2B) tool on creative thinking (primary objective) in adults with psychological disorders. Additionally, the study assesses the B2B effects on energy-related sensations and metabolism, technique adherence, gratefulness and goal-directed activation (secondary objectives) in adults with and without psychological disorders. The observational part of the study primarily aims to investigate the link between psychopathology, intelligence, energy-related sensations and metabolism validating the "c factor mito-bioenergetics" (CMB) model in a sample of adults with and without psychological disorders.

DETAILED DESCRIPTION:
Creativity techniques aim to improve creative thinking and to resolve rigid thinking patterns. They are often recommended and used to generate new insights and perspectives in business and occupational contexts, e.g. to support business development. Despite its successful real-world use, research on the benefits of specific creativity techniques is still in its infancy and it is largely unknown which techniques work best in which contexts.

Most importantly, to the best of the investigators knowledge, (i) specifically designed creativity techniques are not part of any evidence-based psychotherapeutic technique, and (ii) have never been investigated to assist evidence-based psychotherapeutic techniques. Creativity techniques may be helpful in psychotherapy as creative thinking and the generation of new insights and perspectives are believed to be crucial for the efficiency of many psychotherapeutic methods such as cognitive-behavioral therapy and psychodynamic therapy. In addition, it is well-known that people with psychological disorders show less creative thinking, less flexibility and more rigidity in thinking and behavior.

This mixed interventional and observational study has two main aims. The interventional study aims to reveal the effect of a creativity technique - the Brain2Business (B2B) tool - on creative thinking, energy-related sensations and metabolism, technique adherence, gratefulness and goal-directed activation in two different psychotherapeutic techniques (idea generation for pleasurable activities within a behavioral activation therapy (PA-BA) and idea generation for a gratefulness exercise (GE)). As the primary outcome, the acute effect of B2B on creative thinking in adults with a psychological disorder are investigated. As secondary outcomes, the study focuses on the acute B2B effects on energy-related sensations (e.g. tiredness) and metabolism (e.g. heart rate variability) as well as on adherence to the psychotherapeutic techniques, gratefulness and goal-directed activation in adults with and without a psychological disorder.

The B2B tool is a specifically designed creativity technique and depicts a gamified conceptual combination approach. This approach has previously shown to have effects on originality of ideas and it is successfully used in real-world occupational contexts.

The main aim of the observational part of the study is to reveal the relationship between energy-related sensations (e.g., sensations of fatigue and energy), energy metabolism (e.g., heart rate variability, heart rate, core body temperature, skin temperature, blood pressure, cerebral oxygenation), psychopathology, intelligence, and creativity within the newly developed "c factor mito-bioenergetics" (CMB) model. It is a bioenergetic model that links psychopathology and intelligence. The CMB model (i) conceptualizes general cerebral function as the shared variance between intelligence and psychopathology and (ii) assumes that the body's energy metabolism is the biological underpinning of the co-variation between psychopathology and intelligence.

The study will reveal for the first time whether the creativity technique B2B has the potential to assist psychotherapeutic techniques. If the B2B tool efficiently supports creative thinking in psychotherapeutic techniques, clinical trials should follow that compare the psychological effects of a full creativity technique-assisted psychotherapy versus a treatment-as-usual psychotherapy. In addition, the study will evaluate the relation between energy-related sensations and metabolism and validate the CMB model.

ELIGIBILITY:
Inclusion criteria:

* Individuals with and without a diagnosed psychiatric disorder (lifetime or current)

Exclusion criteria:

* Acute suicidality
* Self-reported diagnosed neurological disorders that interfere with the study procedures
* Insufficient German language
* Vulnerable participants (e.g. participants with any indications for an incapability of judgement)
* Caffeine, tobacco consumption and physical activity two hours before the lab-based session starts (only for additional biomarker analyses)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
General creative thinking as assessed with the PTT creativity examination | Measured in the lab-session (time point 4)
  The PTT creativity examination measures general creative thinking in psychotherapeutic techniques (PTT) using a composite measure of a newly developed objective and self-reported creative thinking assessments across two PTT. The composite score is calculated by averaging z-standardized objective and self-reported creative thinking assessments from both PTT. The z-standardized outcome value has a mean of 0 and SD of 1 with a probable range between -3 and +3. Higher scores mean a better outcome. The assessment include the generated ideas (a) for pleasurable activities as a component of behavioral activation (PA-BA) and (b) for a gratefulness exercise (GE). The score will be adjusted for baseline general creative thinking.

SECONDARY OUTCOMES:
Objective creative thinking as assessed with the PTT creativity examination - Objective creativity subscore | Measured in the lab-session (time point 4)
  The objective creativity subscore of the PTT creativity examination is measured with a composite score of fluency, flexibility and originality across different PTT. The composite score is calculated by averaging z-standardized fluency, flexibility, and originality assessments from both PTT. The examination is based on the Torrance Test of Creative Thinking. The z-standardized outcome value has a mean of 0 and SD of 1 with a probable range between -3 and +3. Higher scores mean a better outcome. The score will be adjusted for baseline objective creative thinking.
Self-report creative thinking as assessed with the PTT creativity examination - Self-reported creativity subscore | Measured in the lab-session (time point 4)
  A self-reported creativity composite score about self-generated ideas across different PTT. A newly developed self-report creativity assessment is used with 16 items using a 5-point Likert scale. The sum score ranges from 0 to 64 points. Higher scores mean a better outcome. The score will be adjusted for baseline self-reported creativity (composite of creative self-efficacy and everyday life creativity assessment).
Top 3 creativity evaluation | Measured in the lab-session (time point 4)
  In the Top 3 creativity evaluation a lists of the best three items are rated on creativity by 2 raters. A 5-point Likert scale is used and the sum score ranges from 0 to 15 points. Higher scores mean a better outcome. The score will be adjusted for baseline creative thinking.
PTT creativity examination - Originality subscore | Measured in the lab-session (time point 4)
  A composite measure of objective and self-reported originality. The score will be adjusted for baseline creative thinking.
Eureka moment assessment | Measured in the lab-session (time point 4)
  A newly developed assessment that measures the number of Aha/eureka moments in both psychotherapeutic techniques
Torrance Test of Creative Thinking (TTCT) part II composite score | Measured in the lab-session (time point 4)
  The TTCT part II measures objective creative thinking within the elephant task of the TTCT; 4 minutes; part II). The TTCT composite score is composed of a fluency, flexibility and originality score for the elefphant tasks. The composite score is calculated by averaging z-standardized fluency, flexibility, and originality assessments. The z-standardized outcome value has a mean of 0 and SD of 1 with a probable range between -3 and +3. Higher scores mean a better outcome. The score will be adjusted for baseline objective creative thinking using the TTCT part I without a creativity technique.
Everyday life creativity assessment | Change from pre-test (time point 2) to 1-week-follow-up (time point 5)
  Everyday life creativity is assessed with a newly developed 5-item self-report questionnaire (5-point Likert scale). The sum score ranges from 1 to 5.
Creative self-efficacy | Change from pre-test (time point 2) to 1-week-follow-up (time point 5)
  Creative self-efficacy is assessed with an adapted 6-item creative self-efficacy questionnaire based on two creative self-efficacy questionnaires (5-point Likert scale). The sum score ranges from 6 to 30.
Adherence to behavioral activation (BA) - planned activities | Measured in the lab-session (time point 4)
  Number of planned pleasurable activities during the 5-day diary period
Adherence to behavioral activation (BA) - performed activities | Measured home-based within the 5-day diary period (time point 5)
  Number of performed pleasurable activities during the 5-day diary period.
Adherence to gratefulness exercise (GE) - time | Measured home-based within the 5-day diary period (time point 5)
  The number of minutes people spend in the GE during the 5-day diary period
Adherence to gratefulness exercise (GE) - ideas | Measured home-based within the 5-day diary period (time point 5)
  The number of ideas people created in the GE during the 5-day diary period
Post-acute energy-related sensations as measured with the energy grid | Change within the 5-day diary period measured home-based (time point 5)
  Measured with two energy grid dimensions (wakefulness, sensation of energy) and derived composite scores using mean scores
Bodily sensations of activation/deactivation and lightness/heaviness | Change from pre to post gratefulness exercise in the lab-session (time point 4)
  Measured with the emBody tool
Energy-related metabolism index - acute effects | Change within the lab-session (time point 2 to time point 4)
  A measure validated within the study based on a weighted composite score of all metabolism measures derived from beta coefficients of regression analysis or based on machine learning algorithm.
Energy-related metabolism index - post-acute effects | Change from the lab-session to home-based assessment (time point 2 to time point 5)
  A measure validated within the study based on a weighted composite score of all metabolism measures derived from beta coefficients of regression analysis or based on machine learning algorithm.
Depressive symptoms as assessed Beck Depression Inventory II (BDI II) | Change from pre-test (time point 1) to the last day of the diary period (time point 5)
  The BDI II is a well-validated self-rating questionnaire of depression.
Flow experiences in everyday life as assessed with the Brief Flow Scale (FKS). | Change from pre-test (time point 2) to the last day of the diary period (time point 5)
  The FKS is a validated self-report questionnaire to assess flow experiences
General self-efficacy as assessed with the general self-efficacy brief scale (AKSU) | Change from pre-test (time point 2) to the last day of the diary period (time point 5)
  The general self-efficacy brief scale (AKSU) is a validated self-report questionnaire to assess general self-efficacy
Gratefulness as assessed with the Gratitude questionnaire (GQ-5-G). | Change from pre-test (time point 2) to the last day of the diary period (time point 5)
  The GQ-5-G is a validated self-report questionnaire to assess gratefulness
Creativity exercise experiences | Measured in the lab-session (time point 4)
  A composite measure based on the Game Experience Questionnaire - Core Module, the Energy Grid, and self-developed items. Subscales include challenge - perceived effort, challenge - energy consumption, challenge - perceived task demand, boredomness, competence, pleasant feelings, calmness, sensation of energy, tiredness, match of resources and challenges, self-perceived creativity
Post-creativity exercise experiences as assessed with the Game Experience Questionnaire - post game module | Measured in the lab-session (time point 4)
  A composite measure based on the 4 subscales positive experience, negative experience, tiredness and returning to reality
Acute energy-related sensations | Change within the lab-based session from before the exercises (time point 2) to after each of the exercises (time point 4)
  A composite scores based on the Energy Grid's four dimensions (calmness, pleasant feelings, wakefulness, and sensation of energy).
Goal- and value-based activation | Change from pre-test (time point 2) to the last day of the diary period (time point 5)
  Composite score of the activation subscale of the Behavioral Activation for Depression (BADS) questionnaire and a self-developed value-based activation questionnaire
Physical activity | Change from pre-test (time point 2) to the diary period (time point 5)
  International physical activity questionnaire (IPAQ)
Sleep quality | Change from pre-test (time point 2) to the diary period (time point 5)
  Insomnia scale of the Inventory of Depression and Anxiety Symptoms
Positive/negative experience ratio | Measured at the last day of the diary period (time point 5)
  Ratio of remarkable positive and negative experiences during the 5-day period as measured with a self-developed questionnaire

OTHER OUTCOMES:
Heart rate variability | Change from baseline (time point 2) to exercise tasks (time point 4) within the lab-based session
  Measured with Polar H10 sensor
Core body temperature | Change from baseline (time point 2) to exercise tasks (time point 4) within the lab-based session
  Measured with CORE/CALERAresearch device
Blood oxygenation variability | Change from baseline (time point 2) to exercise tasks (time point 4) within the lab-based session
  SOMNOtouch™ RESP
Variability of beat-to-beat diastolic and systolic blood pressure | Change from baseline (time point 2) to exercise tasks (time point 4) within the lab-based session
  SOMNOtouch™ RESP
24-hour peak-to-peak (maximum-minimum) core body temperature | Change from day 1 to day 3 in the home-based diary period
  Measured with CORE/CALERAresearch device
Respiratory rate | Change from baseline (time point 2) to exercise tasks (time point 4) within the lab-based session
  SOMNOtouch™ RESP
Thoracic/abdominal respiratory ratio | Change from baseline (time point 2) to exercise tasks (time point 4) within the lab-based session
  Measured with SOMNOtouch™ RESP
Cerebral oxygenation | Change from baseline (time point 2) to exercise tasks (time point 4) within the lab-based session
  Sensmart model x-100 NIRS sensors from NONIN
Cerebral oxygenation variability | Change from baseline (time point 2) to exercise tasks (time point 4) within the lab-based session
  Sensmart model x-100 NIRS sensors from NONIN

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Krähenmann, PD, Principal Investigator — Psychiatrische Dienste Thurgau
Locations (1):
- Psychiatric Service Thurgau, Münsterlingen, Thurgau, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
It is not decided because of ethical considerations. If no ethical reasons avoid it, data is planned to be shared.